CLINICAL TRIAL: NCT05342948
Title: Pregnancy Outcome After Secondary Recurrent Pregnancy Loss (sRPL) is Influenced by Sex of the First Born Child and Maternal Carriage of HY-restricting HLA Class II Alleles
Brief Title: Association of HY-restricting HLA Class II Alleles, Sex of Firstborn Child, and Pregnancy Outcome in RPL Patients
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Caroline Nørgaard-Pedersen, Principal investigator, Aalborg University Hospital
Other Study IDs: 2018-5
Record Dates: First submitted 2022-04-07; First posted 2022-04-25 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Maternal immune system; HLA Class II alleles; Habitual Abortion; Immunogenetics; Recurrent Pregnancy Loss
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pRPL: Primary RPL patients: no prior birth ≥22 weeks
- sRPL with a first born boy: Secondary RPL patients: ≥ 1prior birth ≥22 weeks of only boy(s)
- sRPL with a first born girl: Secondary RPL patients: ≥ 1prior birth ≥22 weeks of only girl(s)

SUMMARY:
This cross-sectional and prospective cohort study will investigate if sRPL patients with a first born boy who carry ≥1 HY-restricting (HY-r) HLA class II alleles are associated with a lower chance for a succesful reproductive outcome in first pregnancy after admission compared to sRPL patients with a first born girl carrying ≥1 HY-r HLA class II alleles and women with no HY-r HLA class II alleles and a firstborn boy. Also, the study will compare sRPL patients with a firstborn boy who do not carry a HY-r HLA class II allele with sRPL patients having a firstborn girl and carrying no such alleles.

We hypothesize that sRPL patients with a first born boy compared to sRPL patients with a firstborn girl who carry ≥1 HY-r HLA class II alleles is associated with a negative prognosis, while no association between sex of firstborn child and pregnancy outcome is expected in sRPL carrying no HY-r HLA class II alleles. Neither do we expect an association between pregnancy outcome and carriage of HY-r HLA class II alleles in pRPL patients.

DETAILED DESCRIPTION:
In a Danish cohort (Kolte et al., 2016, Nielsen et al., 2009) the first pregnancy outcome after admission and the long term live birth rate were associated with carriage of known HY-r HLA class II alleles in the sRPL patient with a first born boy, but not in the sRPL with a first born girl. The live birth rate in the first pregnancy after admission and the hazard ratio for live birth on longterm were comparable between sRPL with a first born girl and boy if the sRPL did not carry a HY-r HLA class II allele. In contrast, sRPL after a first born boy had a significant poorer prognosis than sRPL after a first born girl when the patients carried ≥1 HY-r HLA class II allele.

These findings were the first of its kind and it has not been confirmed in other cohorts ever since. In a new Danish cohort from another region of Denmark, this study will examine if these findings can be replicated.

Before data collection, a sample size calculation was performed based on the findings in the former studies (Nielsen et al., 2009; Kolte et al., 2016). These studies differ from the present study, since Nielsen et al. (2009) included HLA DRB3*0301 but not HLA DRB1*07 as a HY-r allele, and Kolte et al.(2016) included HLA DRB3*0301 too and measured the cumulative live birth rate in contrast to first pregnancy outcome measured in the present study. However, the sample size calculation based on weighted calculations on results from these studies is the closest we get a suitable sample size for the present study. The sample size in the present study should consist of at least 88 sRPL patients with a first born boy with maternal HY-r HLA class II allele and 73 sRPL patients with a firstborn boy and no maternal HY-r HLA class II alleles on weighted calculations with an alpha level = 0.05, a power of 80 %, and a inclusion ratio of 1.2 more with than without such HLA carriage. The sample size needed to find difference between women with a firstborn boy vs girl with such HLA carriage was smaller; ie. 48 patients for comparing patients with ≥1 HY-r HLA alleles. As this was the primary aim, this sample size was considered sufficient for the study.

Study inclusion started January 1, 2016, and will end when this sample size is reached.

The anticipated sample size of the pRPL group is 1.2 times the total number of sRPL patients since pRPL normally account for about 55 % of RPL patients. Thus, 180 patients are expected in the pRPL, although this is not taking into account when deciding the timing for final follow-up and data collection.

All RPL patients with ≥3 consecutive pregnancy losses admitted to The Center for Recurrent Pregnancy Loss of Western Denmark who do not have significant uterine malformations, prior birth of children of both sexes, or known chromosomal abnormalities will be included. An obstetric and gynecologic history and a routine blood sample will be obtained on all patients at their first visit according to the ESHRE RPL guideline (2018), on which basis the treatment plan will be decided. The majority of patients have a chromosomal analysis on the patient and her partner and all have a 3D ultrasound, HSU or HSG performed.

Both chemical and clinical pregnancies documented in hospital's or practitioner's records are included, while confirmed molar and ectopic pregnancies are not accounted for.

sRPL is defined as ≥3 pregnancy losses after a pregnancy beyond 22 weeks of gestation while pRPL is defined as ≥3 pregnancy losses with no prior pregnancy beyond 22 weeks of gestation.

Only sRPL with birth of children with same sex prior to RPL will be included in the comparison of sRPL patients with previous boy(s) with sRPL patients with previous girl(s) only.

The primary outcome is the association of reproductive outcome in first pregnancy after admission to our RPL Center with the carriage of HY-restricting HLA class II alleles in the following three groups: sRPL having a first born boy and sRPL having a a girl and also in patients with pRPL.

In addition, we will also explore the prevalence of these HY-restricted HLA class II alleles separately and the sex ratio of births after admission in the three groups.

HLA-DRB1 typing is performed based on genetic analyses of peripheral blood as part of the routine work-up at our clinic.

HY restricted HLA class II alleles in our study is defined as DRB1*01/10 (in strong positive linkage disequilibrium with HLA-DQB1*0501 ); HLA-DRB1*15 and HLA-DRB1*07, which to date have been reported to restrict presentation of HY-antigens.

All data is collected in the RPL clinical database of The RPL Center at Aalborg University Hospital, Denmark (Approval number: 2018-5).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 3 consecutive pregnancy losses before admission

Exclusion Criteria:

* Significant uterine malformation
* Chromosomal abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Among all patients admitted to The Center for Recurrent Pregnancy Loss of Western Denmark from 2016 to 2021 the patients fulfilling study criteria were included and follow up was done continuously until the estimated sample size was reached. The majority of patients were caucasians. Approximately 1/3 of patients were trying to conceive with IVF/ICSI/FER after referral while the remaining 2/3 tried to conceive naturally. About 45% of patients are sPRL patients.
Sampling Method: Non-Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Live birth or prolonged pregnancy in patients with ≥1 HY restricted HLA class II allele | Through study completion, i.e. up to 5 years
  The number of patients with a live birth or prolonged pregnancy (>12 weeks) in first pregnancy after referral with 1-2 HY.-restricted HLA class II allele
Live birth or prolonged pregnancy in patients with 0 HY-restricted HLA class II allele | Through study completion, i.e. up to 5 years
  The number of patients with a live birth or prolonged pregnancy (>12 weeks) in first pregnancy after referral in patients with no HY-restricted HLA class II allele

SECONDARY OUTCOMES:
Maternal prevalence of 0 HY-restricted HLA Class II alleles | Measured on the date of study entry and assessed within 2 weeks for each individual during study completion period, i.e. up to 5 years
  Maternal HY-restricted HLA alleles were considered to be HLA-DRB1*07, -DRB1*15 and DRB1*01/10 (linkage disequilibrium with HLA-DQB1*0501/0502)
Maternal prevalence of ≥1 HY-restricted HLA Class II alleles | Measured on the date of study entry and assessed within 2 weeks for each individual during study completion period, i.e. up to 5 years
  Maternal HY-restricted HLA alleles were considered to be HLA-DRB1*07, -DRB1*15 and DRB1*01/10 (linkage disequilibrium with HLA-DQB1*0501/0502)
Maternal prevalence of HLA DRB1*15 | Measured on the date of study entry and assessed within 2 weeks for each individual during study completion period, i.e. up to 5 years
  One of the three HY restricting HLA class II alleles
Maternal prevalence of HLA DRB1*01 or HLA DRB1*10 | Measured on the date of study entry and assessed within 2 weeks for each individual during study completion period, i.e. up to 5 years
  HLA-DQB1*0501/0502 is one of the three HY restricting HLA class II alleles and this allele is in strong positive linkage disequilibrium with HLA DRB1*01/10 (the total prevalence of patients with ≥1 of these DRB1 alleles)
Maternal prevalence of HLA DRB1*07 | Measured on the date of study entry and assessed within 2 weeks for each individual during study completion period, i.e. up to 5 years
  HLA DRB1*07 is one of the three HY restricting HLA class II alleles
Maternal prevalence of HLA DRB1*03 | Measured on the date of study entry and assessed within 2 weeks for each individual during study completion period, i.e. up to 5 years
  HLA DRB1*03 is one of the HLA class II alleles seen more often than in the background population according to previous studies.
Sex ratio of the children born after RPL | Assessed at the date of study completion, i.e. after 5 years
  Sex ratio of the children born after RPL (i.e. after admission) in each group
Sex ratio of the children born before sRPL | Baseline
  Sex ratio of the children born before RPL diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nørgaard-Pedersen, MD, Principal Investigator — Aalborg University Hospital, Denmark
Locations (1):
- The Centre for Recurrent Pregnancy Loss of Western Denmark, Department of Obstetrics and Gynaecology, Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Background] Kolte AM, Steffensen R, Christiansen OB, Nielsen HS. Maternal HY-restricting HLA class II alleles are associated with poor long-term outcome in recurrent pregnancy loss after a boy. Am J Reprod Immunol. 2016 Nov;76(5):400-405. doi: 10.1111/aji.12561. Epub 2016 Sep 7. PMID 27600856
- [Background] Nielsen HS, Steffensen R, Varming K, Van Halteren AG, Spierings E, Ryder LP, Goulmy E, Christiansen OB. Association of HY-restricting HLA class II alleles with pregnancy outcome in patients with recurrent miscarriage subsequent to a firstborn boy. Hum Mol Genet. 2009 May 1;18(9):1684-91. doi: 10.1093/hmg/ddp077. Epub 2009 Feb 17. PMID 19223392